CLINICAL TRIAL: NCT05878665
Title: Optimizing Low-dose Contrast Media Protocol for Low-kVp Abdominopelvic CT in Suspected Acute Appendicitis
Brief Title: Low-dose Contrast Media for Low-kVp Abdomen CT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bohyun Kim (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Bohyun Kim, Associate professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DLD-001
Record Dates: First submitted 2023-03-23; First posted 2023-05-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Appendicitis Acute
Keywords: acute appendicitis; acute abdomen; CT
MeSH Terms: conditions — Appendicitis; Abdomen, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Double low-dose CT (Experimental): Weight-adjusted low-dose contrast media paired with low-radiation dose abdomen CT
  Interventions: Diagnostic Test: Weight-adjusted low-dose contrast media paired with low-radiation dose abdomen CT

INTERVENTIONS:
Diagnostic Test: Weight-adjusted low-dose contrast media paired with low-radiation dose abdomen CT — The investigators are aiming for a 10% reduction in iodine dosage at 10 kVp reduction in CT radiation. Routine iodine dosing is 0.521 g I/kg at 120 kVp. Therefore, at 90 kVp, a 30% reduction in iodine dosing is expected, which is 0.365 g I/kg. At 100 kVp, the iodine dosage is reduced to 0.417 g I/kg, which is a 20% reduction. The kVp value is automatically selected by the CT device according to the body habitus, which is a clinical routine.

SUMMARY:
The purpose of this clinical study is to test the performance of low radiation dose abdominal CT combined with low dose contrast media for the diagnosis of acute appendicitis in young patients. The main questions to be answered are:

1, Can low-dose contrast media paired with low-dose radiation CT of the abdomen provide acceptable diagnostic accuracy in acute appendicitis? 2. How much radiation dose can be saved by using low radiation dose abdominal CT in combination with low dose contrast media?

ELIGIBILITY:
Inclusion criteria:

* Patients in the emergency department with suspected acute appendicitis based on clinical examination
* Patients scheduled for contrast-enhanced CT of the abdomen and pelvis for diagnosis of suspected acute appendicitis.

Exclusion criteria:

* Patients who decline to participate
* Contraindications to contrast-enhanced CT (eGFR < 30 mL/min/173 m^2 or pregnant)
* BMI >= 30.

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 292 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy for acute appendicitis | For operated patients, postop. period (up to 1 month); If non-operated, at 6 months-FU
  The primary outcome of the study is the diagnostic accuracy of double low-dose CT for acute appendicitis in young adults with suspected acute appendicitis. Based on the CT findings, a three-tiered diagnosis of appendicitis will be given (no appendicitis, uncomplicated appendicitis, or complicated appendicitis). In the case of no appendicitis, a possible alternative diagnosis is given. The reference standard for appendicitis is operative findings and surgical pathology reports. In nonoperative cases, sequential radiologic evaluation, clinical follow-up, and the judgment of the attending physician will conclude the diagnosis. Specifically, if the patient is not treated for recurrent symptoms within 6 months, the radiologic diagnosis of CT findings is considered valid. The diagnostic accuracy for acute appendicitis is true positive for acute appendicitis and true negative for acute appendicitis divided by all participants.

CONTACTS AND LOCATIONS:
Overall Officials: Bohyun Kim, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No